CLINICAL TRIAL: NCT01561326
Title: Facilitating Follow-Up Adherence for Abnormal Pap Smears
Acronym: TC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Temple University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB04802; R01CA104979 (NIH)
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Uterine Cervical Neoplasms
Keywords: cervical cancer; follow-up; Pap test; Medical management; Colposcopy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive-affective barriers counseling delivered by phone (Experimental): Standard care plus cognitive-affective barriers counseling delivered by phone , i.e., culturally-relevant/sensitive barrier-specific messages drawn from a pre-developed library designed to counsel individuals regarding their specific barriers to adherence
  Interventions: Behavioral: Cognitive-affective barriers counseling
- cognitive-affective barriers counseling via brochure (Experimental): Standard care plus cognitive-affective barriers counseling delivered via mail-home print material
  Interventions: Behavioral: Cognitive-affective barriers counseling via brochure
- standard care (Active Comparator): Cognitive-affective barriers (CAB) assessment delivered via phone; receipt of a notification letter from physician regarding abnormal Pap test result, need to undergo colposcopy, appointment date and clinic contact numbers; telephone confirmation and post-card appointment reminder
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: Cognitive-affective barriers counseling — Culturally-relevant/sensitive barrier-specific messages drawn from a pre-developed library designed to counsel individuals regarding their specific barriers to adherence, e.g., by increasing risk-related knowledge, providing accurate outcome and self-efficacy expectancies, addressing health-related values and goals, moderating risk-related affect, or offering active plans and strategies to assist with self-regulation
  Arms: Cognitive-affective barriers counseling delivered by phone
Behavioral: Cognitive-affective barriers counseling via brochure — Culturally-relevant/sensitive barrier-specific messages drawn from a pre-developed library designed to counsel individuals regarding their specific barriers to adherence via brochure, e.g., by increasing risk-related knowledge, providing accurate outcome and self-efficacy expectancies, addressing health-related values and goals, moderating risk-related affect, or offering active plans and strategies to assist with self-regulation
  Arms: cognitive-affective barriers counseling via brochure
Behavioral: standard care — Cognitive-affective barriers (CAB) assessment delivered via phone; receipt of a notification letter from physician regarding abnormal Pap test result, need to undergo colposcopy, appointment date and clinic contact numbers; telephone confirmation and post-card appointment reminder
  Arms: standard care

SUMMARY:
Objective: Previous studies have suggested that psycho-educational interventions delivered by telephone improve adherence to initial colposcopy after an abnormal Pap smear. To further explore strategies for enhanced follow-up to medical care recommendations, we studied the impact of a theory-guided cognitive-affective barriers counseling intervention, delivered at 2-4 weeks before the colposcopy appointment, for inner city women. The comprehensive telephone barriers intervention was compared to an enhanced comparison group and a group that received tailored print materials.

Methods: Participants (N = 211) were recruited through a colposcopy clinic and randomly assigned to: 1) telephone assessment of barriers to follow up adherence recommendations combined with tailored telephone barriers counseling; 2) telephone assessment combined with tailored barriers print brochure; or 3) telephone assessment with no barriers counseling. Participants were assessed at baseline, 1-week, 9 and 15 months post-colposcopy.

DETAILED DESCRIPTION:
Objective: Previous studies have shown that theory-based, tailored telephone barriers counseling significantly improves adherence to a colposcopy appointment after an abnormal pap smear result among low-income, minority women. This study built on these research findings and explored the efficacy of a state-of-the-science telephone counseling intervention utilizing a more rigorous study design. This enhanced counseling intervention was tailored to individual's distinctive cognitive-affective barriers profile, as assessed by the Cognitive-Social Health Information Processing (C-SHIP) model-guided barriers assessment tool, and with counseling messages targeted to all five domains of individual's barriers to adherence. In addition, the current study design was improved in two ways. First, the comparison group in this current study was an enhanced one that received a notification letter, assessment of cognitive-affective barriers by telephone, and a telephone appointment reminder. Second, this study had a longer follow-up period to allow testing of the intervention effect beyond initial colposcopy adherence. The participants were followed for 15 months post-colposcopy so that participants' adherence to medical follow-up recommendations (if any) within the 12 months after initial colposcopy can be collected and studied. Adherence to medical follow-up at 6 months and 12 months was measured at 9 months and 15 months, respectively, to allow 3 months for rescheduling, attending, and recording of the appointment. Overall, this study tested whether an enhanced tailored telephone barriers counseling intervention improve adherence to medical follow-up after abnormal pap smear among low-income, minority women.

Methods:

METHODS Participants (211) were randomized to the following baseline conditions: a) standard care (SC), i.e., a cognitive-affective barriers (CAB) assessment delivered via phone, receipt of a notification letter from physician regarding abnormal Pap test result and need to undergo colposcopy, and also including appointment date and clinic contact numbers, plus telephone confirmation and post-card appointment reminder; b) SC plus CAB counseling delivered by phone (CAB-C -T), i.e., culturally-relevant/sensitive barrier-specific messages drawn from a pre-developed library designed to counsel individuals regarding their specific barriers to adherence, e.g., by increasing risk-related knowledge, providing accurate outcome and self-efficacy expectancies, addressing health-related values and goals, moderating risk-related affect, or offering active plans and strategies to assist with self-regulation; c) SC plus CAB counseling delivered via Mail-Home Print Material (CAB-C-P), which included exactly the same applicable messages as were delivered by phone, but in print form. The tailoring of messages to a participant's cognitive-affective barriers profile was based on the two barriers in each of the five Cognitive-Social Health Information Processing (C-SHIP) categories (a total of 10 messages) that she rated most important on a five-point scale. There were 23 cognitive-affective adherence barriers grouped into the following C-SHIP categories: 1) risk-related encodings/perceptions (i.e., purpose of colposcopy, presence and progression of HPV-related disease); 2) risk-related expectancies and beliefs (i.e., confidence in ability to keep appointment, fatalistic beliefs about cancer); 3) risk-related values and goals (i.e., maintaining modesty, importance of having children); 4) risk-related affect (i.e., worries about necessary procedures and/or progression of disease, concerns regarding fertility); and 5) risk-related self-regulation (i.e., remembering appointment, overcoming child-care or work-related conflicts, transportation difficulties, ability to manage any negative risk-related affect). With regard to assessments, they were conducted at the following time points: baseline, and 1-week, 9-month, and 15-month post-colposcopy and included the following: the CAB assessment; background variables, including demographic (e.g., gender, age, ethnicity, education, marital and employment status, household income, number of children); medical and screening history (e.g., cancer diagnosis, previous Pap smears and frequency; breast exams (self and clinical); mammograms and abnormal results; results of the index colposcopy and physician recommendations from medical records; a potential moderating dispositional variable, attentional style (Monitoring-Blunting Style Scale); potential mediating variables, including affective variables (Spielberger State-Trait Anxiety Inventory, the Center for Epidemiological Studies-Depression Scale), and cognitive-affective process variables (knowledge, risk perceptions, expectancies and beliefs, affect, values and goals, regulatory skills); outcome variables, including adherence to initial diagnostic colposcopy and to 6- and 12-months colposcopically-based follow-up diagnostic and medical management recommendations, and an intervention evaluation. All assessments used scales developed in previous research, except the Powe Fatalism Inventory used to assess fatalism and the Revised Impact of Events Scale used to assess affect (i.e., stress-related intrusive and avoidant thoughts). Assessed at baseline were background variables (except medical recommendations), the moderating variable, and all mediating variables. The cognitive-affective barriers were assessed only at baseline. Assessed at 1-week post-colposcopy and at the 9-month and 15 month follow-ups were all mediating variables (except the cognitive-affect barriers) and outcome variables. The medical recommendations were assessed only at the 1-week post-colposcopy. Medical history was also re-assessed at the 15-month follow-up relating to the interim period from baseline.

ELIGIBILITY:
Inclusion Criteria:

* women 18 years old or older
* have recently received an abnormal Pap smear indicative of oncogenic HPV
* have been referred for initial colposcopic evaluation at the Women's Care Center at Temple University Hospital
* able to communicate with ease in English

Exclusion Criteria:

* unable to communicate readily in English
* do not have access to a telephone
* have a history of any malignancy
* display current evidence of positive invasive carcinoma of the cervix
* display presence of another life-threatening medical condition
* show evidence of dementia
* prior participation in research study
* HIV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2005-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Adherence to diagnostic colposcopy appointment | 1-week Post-Colposcopy
  Adherence to initial diagnostic colposcopy will be assessed for each participant through tracking of clinic reports/patient medical records immediately post-colposcopy. Adherence will be measured dichotomously with patients who attend their initial appointment or who cancel their initial colposcopy appointment but reschedule within one month of their original date deemed adherent and eligible for follow-up assessments.

SECONDARY OUTCOMES:
Adherence to long-term follow-up medical recommendations | 9- and 15-months post-index appointment
  Adherence to 6- and 12-months colposcopically-directed recommendations and medical management over time will be assessed through medical chart review, as well as self-report, at 9- and 15-months post-index appointment. A 3-month grace period was selected to accommodate any clinic-based rescheduling and/or cancellation of appointments for procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M. Miller-Halegoua, Ph.D., Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States